CLINICAL TRIAL: NCT03170791
Title: Feasibility and Acceptability of Transcutaneous Vagal Nerve Stimulation in Recovery of Upper Limb Function Post Stroke
Brief Title: Noninvasive Vagal Nerve Stimulation for Arm Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STH19008
Record Dates: First submitted 2017-05-12; First posted 2017-05-31 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vagal nerve stimulation intervention (Experimental): All participants consented to the study will undergo an exercise session using equipment such as pedals and cylinders to facilitate activity. During the exercise session the therapist will press a switch to trigger a run of vagal nerve stimulation in time with the patient's activity. Patients will be videoed during the therapy sessions to allow researchers to retrospectively count the number and type of repetitive movements successfully performed. At the end of the exercises, the stimulator clip will be removed from the patient's ear and cleaned with an alcohol disinfectant wipe ready for next use.
  Interventions: Device: vagal nerve stimulation intervention

INTERVENTIONS:
Device: vagal nerve stimulation intervention — During exercise sessions the therapist will the therapist will press a switch to trigger a run of vagal nerve stimulation in time with the patient's activity. No further activity involved.

SUMMARY:
This study will find out whether electrical stimulation of a nerve called the "vagus" nerve is acceptable for patients undergoing physiotherapy for arm weakness after a stroke. 20 patients will be recruited if they had a stroke between 4 and 48 months previously and have been left with reduced function in the affected arm. Patients will receive 3 sessions of physiotherapy per week for 6 weeks. Each session will last 1 hour during which the patient will be asked to perform specific movements e.g. shuffling cards, reaching for a shelf. With each arm movement the therapist will turn on a stimulator which is worn clipped to the patients ear. This will deliver a short burst of electricity creating a mild tingling sensation.

At the end of the session, the stimulator will be removed and the patient will be asked to rate the level of any discomfort or fatigue they experienced as well as any other side effects. The therapist will also record whether the stimulator device interfered with the therapy in any way. A heart tracing will be performed at each visit to check the heart rhythm. At the start and end of the 6 week course of physiotherapy, patients arm weakness and level of arm function will be assessed, as well as their general levels of fatigue, mood and quality of life. These will be reassessed at 1 month and 6 months after the course of physiotherapy has ended. The investigators will also interview patients to establish how they found the treatment itself. If the vagal nerve stimulation combined with physiotherapy is acceptable to patients and therapists and there are no safety concerns, the investigators will plan a larger trial of this treatment in stroke patients.

DETAILED DESCRIPTION:
This study will find out whether electrical stimulation of a nerve called the "vagus" nerve is acceptable for patients undergoing physiotherapy for arm weakness after a stroke. 20 patients will be recruited if they had a stroke between 4 and 48 months previously and have been left with reduced function in the affected arm. Patients will receive 3 sessions of physiotherapy per week for 6 weeks. Each session will last 1 hour during which the patient will be asked to perform specific movements e.g. shuffling cards, reaching for a shelf. With each arm movement the therapist will turn on a stimulator which is worn clipped to the patients ear. This will deliver a short burst of electricity creating a mild tingling sensation.

At the first visit to the Clinical research Facility, the researcher will check that the patient is still happy to take part. Then, some information about the patient e.g. age, sex, date of stroke, risk factors for stroke will be recorded. Next, the therapist will assess how much existing strength and function the patient has in the arm affected by their stroke using a variety of rating scales. Some brief questionnaires will also be used to measure the patients levels of depression, anxiety, fatigue, quality of life and levels of independence.

These initial assessments will take approximately one hour and will be conducted at the first visit, before the exercises commence. Next the research physiotherapist will clean the patients ear using an alcohol wipe then apply the vagal nerve stimulator clip to part of the ear. The stimulator will be set to deliver a burst of electricity which the patient will feel as a tingling sensation that is not uncomfortable.

The exercise session will then commence with a five minute warmup consisting of whole arm movements using equipment such as pedals and cylinders to facilitate activity. The patient will then be asked to perform a range of practical tasks using their weak arm e.g.turning cards, moving objects of various shapes and sizes, opening and closing bottles and bilateral activities such as lifting objects with both hands. The exercise regime will aim to incorporate 300- 400 such arm movements and will take approximately one hour.

During the exercises, the therapist will press a switch to trigger a run of vagal nerve stimulation in time with the patient's activity. Patients will be videoed during the therapy sessions to allow researchers to retrospectively count the number and type of repetitive movements successfully performed. At the end of the exercises, the stimulator clip will be removed from the patient's ear and cleaned with an alcohol disinfectant wipe ready for next use. After each therapy session, patients will be asked to document on scale of 05 how much they experienced skin reddening, irritation, nausea, dizziness, and headache. Patients will be asked to rate their level of discomfort and fatigue arising from the session using a 05 scale.

Patients will also be given a diary to take home to record details of any physiotherapy sessions they undergo outside the study (including any exercise they do at home) and any new symptoms that may arise. They will be asked to bring this diary to the remaining sessions. The patient will undergo 3 of these exercise sessions per week for 6 weeks (i.e. 18 exercise sessions altogether). The remaining 17 session will begin with application of the stimulator clip and the warm up as detailed above. At the end of the final exercise session, the scales used to measure arm strength and function, mood, fatigue and quality of life will be repeated.

Patients will then return to the Clinical Research Facility after 1 month and after 6 months to have their arm function tests repeated and to reassess their mood, quality of life and fatigue. No exercise will be performed at these last 2 visits.

The patients who receive physiotherapy during October- December 2015 will be invited to take part in a separate interview with the MSc student who has been delivering their physiotherapy. This will take place at a mutually convenient time at the Clinical Research Facility. During that interview, the patient will be asked how they found the treatment, whether there were any problems and whether it was what they expected. These interviews will be tape recorded so that the student can listen to the tapes and analyse what the patients have said.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age >18) patients will be invited to take part if they suffered a stroke between 3 months and 2 years previously
* The patient must have moderate to severe upper limb limitation (Upper Extremity Fugl-Meyer score 2050) due to the stroke
* Patients must have a minimum of 10 degrees of active wrist extension, 10 degrees of active thumb abduction/extension and 10 degrees active extension in at least 2 additional digits.

Exclusion Criteria:

* Other significant impairment of upper limb e.g. frozen shoulder
* Other diagnosis likely to interfere with rehabilitation/outcome assessments e.g. registered blind
* Patients with insufficient language skills to give informed consent and provide feedback both during the therapy sessions and in a semi structured interview.
* Severe cardiovascular disease or pathological ECG at baseline
* Patients participating in another rehabilitation trial
* Pregnant or trying to get pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Patient Safety as measured by patient reported adverse events | 12 months
  Patient safety will be assessed with ECG recordings at each therapy visit, by review of the diary of side effects and investigation of any adverse events.

SECONDARY OUTCOMES:
Acceptability of study | 12 months
  Patient acceptability will be assessed by patient feedback during the qualitative interviews
Feasibility of study as measured by number of completed therapy sessions | 12 months
  Study feasibility will be assessed by review of number of therapy sessions fully completed and the number of repetitive movements achieved in one hour

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Majid, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no individual participant data will be shared